CLINICAL TRIAL: NCT00200096
Title: Acupuncture for the Treatment of Chronic Post-Chemotherapy Fatigue: A Randomized, Phase III Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Gary Deng, MD,PhD, Memorial Sloan Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 04-081
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Cancer
Keywords: Cancer; Fatigue
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Acupuncture and questionnaires
  Interventions: Procedure: Acupuncture and questionnaires
- 2 (Sham Comparator): placebo acupuncture and questionnaires
  Interventions: Procedure: placebo acupuncture

INTERVENTIONS:
Procedure: Acupuncture and questionnaires — Acupuncture once weekly for six weeks Brief Fatigue Inventory, Hospital Anxiety and Depression Scale, Functional Assessment of Cancer Treatment scale. Patients will repeat the BFI and FACT-G at seven and eight weeks after randomization, approximately one and two weeks after their final treatment. HADS will be repeated at week seven. At the end of the study, patients will be asked to state whether they were thought they on true or placebo acupuncture and why.
  On the day of the final session of acupuncture treatment (approximately day 35), blood samples will be collected and tested for hemoglobin, thyroid function tests, as described in pretreatment evaluation. The results will be designated "posttreatment" values. Actigraphic monitoring will be conducted in week seven. Patients will be asked to wear the device for seven days just like during baseline evaluation.
  Arms: 1
Procedure: placebo acupuncture — During the placebo phase, placebo acupuncture needles (68) will be applied a few mm away from the points. The placebo acupuncture needle is a blunt tipped needle that moves up inside its handle. However, the needle does not penetrate the skin and instead moves upward inside the handle. Needles will be applied after sterile swabbing of the skin and kept in place for 20 minutes in both group.Patients in the placebo group will be offered true acupuncture after receipt of the week seven and eight fatigue diaries.
  Patients will complete the BFI, HADS and FACT-G at baseline, approximately two weeks before randomization and their first treatment. The BFI and FACT-G will be repeated after seven days, that is, one week before randomization. The use of repeat measurement decreases intrapatient variability and hence increases the precision of the baseline measure.
  Arms: 2

SUMMARY:
In a previous study, we found that acupuncture may decrease fatigue. The aim of this study is to determine whether acupuncture is helpful in reducing fatigue in cancer patients treated with chemotherapy. We will also study how fatigue, quality of life, mood, level of physical activity. This study will involve about 88 patients.

DETAILED DESCRIPTION:
Primary objective:

To determine whether acupuncture reduces chronic fatigue after chemotherapy more effectively than placebo

Secondary objectives:

1. To examine the long-term effects of acupuncture treatment on fatigue
2. To examine predictors of response to acupuncture treatment in terms of baseline symptoms, hemoglobin, age, sex, time since chemotherapy and concurrent treatment
3. To examine the effect of acupuncture on levels of physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 64 diagnosed with a malignancy (solid tumor or hematologic malignancy). We are excluding children primarily because fatigue in children is assessed differently from adults (56). Moreover, as children constitute only about 5% of the cancer population and as post-chemotherapy fatigue appears to be relatively rare in children (57), we would expect little if any accrual from the pediatric population. Patients aged 65 and over are excluded for likely non-response, as described under preliminary data.
* Patients must have received chemotherapy
* Patients must complain of fatigue following chemotherapy but not prior to chemotherapy
* At least 60 days must have elapsed between the last chemotherapy infusion and completion of the first baseline questionnaire. Acute chemotherapy related fatigue typically lasts two to three weeks at most (58). Patients with fatigue at 60 days can therefore be considered to be chronic cases.
* Mean baseline fatigue as measured by the Brief Fatigue Inventory (BFI) must be four or above. A score of four on the BFI is considered the threshold between "mild" and "moderate" symptoms (18).

Exclusion Criteria:

* Anemia, defined as Hb<9 or active treatment for anemia. Iron supplementation is allowed as long as the dose has been stable for at least six weeks. Anemia is excluded as a major treatable cause of fatigue.
* Platelets less than 50,000/microliter or an Absolute Neutrophil Count less than 1,000/microliter. Patients with low platelets or neutrophils are at the risk of bleeding or infection, respectively.
* Baseline depression score on the Hospital Anxiety and Depression Scale of 11 or above, indicating clinical depression. Patients excluded for depression will be referred for appropriate psychiatric evaluation. Depression is excluded as a treatable cause of fatigue.
* Thyroid disorder, defined as either thyroid stimulating hormone or free T4 out of normal range, is excluded as it is a possible cause of fatigue unrelated to cancer therapy.
* Surgery under general anesthesia; immunotherapy; radiotherapy; or initiation of hormonal therapy within the three weeks prior to enrollment.
* Acupuncture in the previous six weeks.
* Change in use of any of the following drugs in the prior three weeks: opiates, anti-depressants (other than selective serotonin reuptake inhibitors [SSRIs]) / anxiolytics; OR change in use of SSRIs in the prior six weeks. "Change in use" is defined as initiation or cessation of treatment, or change in prescribed dose or regimen: changes in actual amounts of PRN medication taken are allowed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2004-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine whether acupuncture reduces chronic fatigue after chemotherapy more effectively than placebo | six weeks

SECONDARY OUTCOMES:
To examine the long-term effects of acupuncture treatment on fatigue | six months
To examine predictors of response to acupuncture treatment in terms of baseline symptoms, hemoglobin, age, sex, time since chemotherapy and concurrent treatment | six months
To examine the effect of acupuncture on levels of physical activity and quality of life. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://mskcc.org